CLINICAL TRIAL: NCT07192289
Title: Using Platelet-rich Fibrin in Regenerative Endodontic Treatment in Mature Permanent Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: Odonto-Maxillo Facial Hospital in Ho Chi Minh City (Unknown)
Responsible Party: Principal Investigator, Tran Thi Tuong Vi, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3787/QĐ-ĐHYD
Record Dates: First submitted 2025-09-07; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Apical Periodontitis; Necrosis of Pulp; Acute Apical Periodontitis of Pulpal Origin; Periapical Abscess
Keywords: PRF; regenerative endodontic treatment; mature permanent treatment
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Abscess | interventions — proliferation regulatory factors, human urine; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Control Group - Blood clot method for regenerative endodontics. Experimental Group 1 - Regenerative endodontics using advanced platelet-rich fibrin (A-PRF+).
  Experimental Group 2 - Regenerative endodontics using injectable platelet-rich fibrin (i-PRF).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Using advanced platelet-rich fibrin (A-PRF+) or injectable platelet-rich fibrin (i-PRF) in regenerative endodontic treatment in mature permanent teeth. — After obtaining informed consent, the study will be conducted over 2 appointments, 2-4 weeks apart.
  The first appointment will focus on infection control and inflammation reduction. The canal will be instrumented with a single-file system. The canal will be then irrigated sequentially with 3% sodium hypochlorite (NaOCl), saline, and 17% ethylenediaminetetraacetic Acid (EDTA) to ensure thorough disinfection. Finally, a temporary filling of Glass Ionomer Cement will be placed over an intracanal dressing of calcium hydroxide.
  At the second appointment, the final treatment will be performed based on the patient's group:
  Control Group - Blood clot method for regenerative endodontics. Experimental Group 1 - Regenerative endodontics using advanced platelet-rich fibrin (A-PRF+).
  Experimental Group 2 - Regenerative endodontics using injectable platelet-rich fibrin (i-PRF).
  All three groups will be then sealed with mineral trioxide aggregate (MTA) and a final composite resin filling.
  Other Names: PRF in regenerative endodontic treatment

SUMMARY:
This study aims to evaluate the antibacterial effects of injectable platelet-rich fibrin (i-PRF) in vitro, and to assess the clinical and radiographic outcomes of using advanced platelet-rich fibrin (A-PRF+) and i-PRF in regenerative endodontic treatment of mature permanent teeth with necrotic pulp. The study will compare the effectiveness of PRF-based treatment with conventional blood clot-based regenerative endodontics.

DETAILED DESCRIPTION:
This study aims to evaluate the antibacterial effects of injectable platelet-rich fibrin (i-PRF) in vitro, and to assess the clinical and radiographic outcomes of using advanced platelet-rich fibrin (A-PRF+) and i-PRF in regenerative endodontic treatment of mature permanent teeth (single-rooted teeth with necrotic pulp, with or without periapical pathology). The study will compare the effectiveness of PRF-based treatment with conventional blood clot-based regenerative endodontics.

ELIGIBILITY:
Inclusion Criteria:

Participants had a single-rooted tooth with necrotic pulp (negative response to electric pulp testing), with or without periapical pathology (acute apical periodontitis of pulpal origin, chronic periapical periodontitis, periapical abscess with sinus, periapical abscess without sinus), and gave their consent to participate in the study.

Exclusion Criteria: Study samples will be excluded if any of the following criteria are met:

* The tooth has had previous endodontic treatment.
* The root apex is not fully developed, or there is root resorption/cracking/fracture.
* The tooth has severe tooth loss and is indicated for extraction, or is indicated for restoration with a post or cast core after endodontic treatment.
* The root canal is calcified.
* The root canal curvature is greater than 25º.
* The tooth has a periapical cyst or is associated with a jawbone cyst.
* The tooth has a periodontal pocket deeper than 4 mm.
* The tooth has no occlusal contact.
* The patient is pregnant.
* The patient has diabetes or HIV or other immunocompromised conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment | 1 month, 3 months, 6 months, 9 months, 12 months.
  * Clinical success: Absence of all the following symptoms (swelling, sinus tract, pain on percussion/bite, tooth mobility, and positive pulp sensibility).
  * Clinical failure: Presence of any one of the above symptoms.
Radiographic assessment | 1 month, 3 months, 6 months, 9 months, 12 months
  * Radiographic success: Absence or reduction of periapical pathology, measured by change in lesion size on periapical radiographs/CBCT.
  * Radiographic failure: Persistence or progression of periapical pathology, measured by change in lesion size on periapical radiographs/CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Odonto-Maxillo-Facial Hospital and University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
To ensure patient data confidentiality, I do not intend to share the research data with other researchers.